CLINICAL TRIAL: NCT07322679
Title: Effects of Dihydroberberine Supplementation on Body Composition, Glycemic Control, Energy Levels, Appetite, and Mood in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial
Brief Title: Dihydroberberine Effects on Body Composition and Metabolic Health in Healthy Adults
Acronym: DHB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Nutrabuilding Bio-tech Co., Ltd. (Other)
Collaborators: Biofortis, Merieux NutriSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NNBHCS-BIO-2513
Record Dates: First submitted 2025-12-12; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Health Adult Subjects
Keywords: Glucovantage®; DHB; Dihydroberberine; Body Composition; Glycemic Control; Energy Levels; Appetite; Mood; metabolism; Blood glucose; Body weight management; Waist circumference; Hip circumference; Leptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo （Microcrystalline Cellulose）
- Dihydroberberine（DHB） (Experimental)
  Interventions: Dietary Supplement: Dihydroberberine（DHB）

INTERVENTIONS:
Dietary Supplement: Placebo （Microcrystalline Cellulose） — Participants will take 4 placebo capsules daily for 12 consecutive weeks, with 2 capsules taken in the morning and 2 in the evening. Each capsule contains 200 mg of microcrystalline cellulose, an inert substance used as an inactive control.
  Arms: Placebo
Dietary Supplement: Dihydroberberine（DHB） — Participants will take 4 capsules daily (each containing 100 mg dihydroberberine [DHB] and 100 mg microcrystalline cellulose) orally for 12 consecutive weeks, with 2 capsules taken in the morning and 2 in the evening. The total daily dose of DHB is 400 mg.
  Arms: Dihydroberberine（DHB）

SUMMARY:
The goal of this clinical trial is to evaluate whether dihydroberberine (DHB) supplementation can improve body composition, blood sugar control, energy levels, appetite, and mood in healthy adults with overweight or mild obesity. The study focuses on men and women aged 35-55 years with a BMI between 27.0 and 33.0 kg/m².

The main questions it aims to answer are:

Does daily DHB supplementation lead to greater reductions in body weight over 12 weeks compared to placebo? Does DHB improve glycemic responses, appetite regulation, energy levels, and mood, both acutely (short-term) and chronically (over 12 weeks)?

Researchers will compare two groups-one receiving DHB (400 mg/day) and the other receiving a placebo-administered as two capsules twice daily for 12 weeks. Participants will:

Attend three in-clinic visits over approximately 14 weeks (including screening, baseline, and week 12 visits) Undergo mixed-meal tolerance tests (MTTs) to assess glucose metabolism, appetite, and energy levels Complete body composition assessments (including DXA scans), blood tests (e.g., glucose, insulin, HbA1c), and mood questionnaires (POMS-2) Be monitored for safety throughout the study

ELIGIBILITY:
Inclusion Criteria:

* 35 - 55 years of age (inclusive) at visit 1.
* BMI ≥ 27.0 - ≤ 33.0 kg/m2.
* Participant has a score of 7 - 10 on the Vein Access Scale Assessment at visit 1.
* Non-user or former user (daily use; cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1, and has no plans to begin use during the study period.
* Non-habitual users (i.e., daily or almost daily) of marijuana or hemp products, including CBD/THC products, and willing to abstain from use throughout the study period (topical creams/lotions are allowed).
* Willing to use personal smart phone with operating system capable of downloading and operating study applications (e.g., FitBit, smart scale, activity watch, etc).
* Willing to adhere to all study procedures, including lifestyle considerations (see section 6.3), and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

* Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan/vegetarian) at the discretion of the Clinical Investigator.
* Individuals undergoing moderate-to-intense activity (e.g., sports/exercise ≥ 5h/wk).
* Recent weight changes (>4.5 kg ≤ 90 d of visit 1), or current/planned engagement in a weight change program (e.g., weight loss or muscle gain) outside of the researcher-instructed, self-directed Lifestyle Intervention throughout the study period.
* Abnormal laboratory test results of clinical significance at visit 1, at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to visit 2, for subjects with abnormal laboratory test results.
* Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions that are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
* Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies).
* Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg. Stable use (no initiation or change in dose ≤ 90 d of visit 1) of FDA-approved medications for hypertension is allowed.
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Signs or symptoms of an active infection of clinical relevance ≤ 5 d of visit 1. The visit may be rescheduled once all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 d prior to visit 1.
* Recent use (≤ 6 mo of visit 1) of any prescription anti-hyperglycemic/weight loss medication. This includes, but is not limited to: metformin, insulin, DPP-4 inhibitors, SGLT-2 inhibitors, GLP-1 agonist, GIP agonists, Pioglitazone and Sulfonylureas.
* Use of any dietary supplement, other than conventional once-daily multivitamin/mineral supplements (within limits of the DRI) ≤ 14 d of visit 1 and throughout the study.
* Recent history (≤ 12 months visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Unstable use (change in dose) of any other prescription medications ≤ 90 d of visit 1, except for medications used PRN (e.g., asthma inhalers, non-drowsy seasonal allergy medications, etc.)
* Antibiotic use ≤ 90 d of visit 1 and throughout the study period.
* Regular use (≥ 3 days/week ≤ 30 d of visit 1) of anti-inflammatory medications (e.g., NSAIDs) and throughout the study period.
* Recent use of oral or injectable steroids, or topical or inhaled steroids (≥ 1500 µg/d) within 30 d of visit 1 and throughout the study period.
* Exposure to any non-registered drug product ≤ 30 d prior to visit 1.
* Diagnosed with major affective disorder, or other psychiatric disorder, that required hospitalization ≤ 12 months prior to visit 1.
* Recent (≤ 90 d of visit 1) endoscopy and/or colonoscopy procedure.
* Major trauma or any other surgical event ≤ 30 d of visit 1.
* Currently scheduled, or planning to schedule, an elective surgical procedure during the study.
* Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Women who become pregnant during the study will be discontinued.

General safety related criteria

* Known sensitivity, intolerability, or allergy to any of the study products or study foods.
* Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, and comply with the study protocol, which might confound the interpretation of the study results, or put the participant at undue risk.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Body weight will be measured in-clinic at Baseline (Visit 2, Week 0, Day 1) and End of Study (Visit 3, Week 12, Day 84) using a calibrated digital scale under standardized conditions (fasted, light clothing, no shoes).

SECONDARY OUTCOMES:
Plasma Glucose Positive Incremental Area Under the Curve (piAUC) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Positive incremental Area Under the Curve (piAUC0-120min) of plasma glucose following a Mixed-meal Tolerance Test (MTT) after a single dose of study product.
Plasma Glucose Maximum Concentration (Cmax) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Maximum concentration (Cmax) of plasma glucose following a Mixed-meal Tolerance Test (MTT) after a single dose of study product.
Plasma Glucose Time to Maximum Concentration (Tmax) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Time to maximum concentration (Tmax) of plasma glucose following a Mixed-meal Tolerance Test (MTT) after a single dose of study product.
Composite Appetite Score Net Incremental Area Under the Curve (niAUC) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Net incremental Area Under the Curve (niAUC0-120min) for the Composite Appetite Score following a Mixed-meal Tolerance Test (MTT) after a single dose of study product.
Net Incremental Area Under the Curve (niAUC0-120min) for Individual Appetite Visual Analog Scale (VAS) Ratings | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Net incremental area under the curve (niAUC) from 0 to 120 minutes for individual appetite-related sensations measured using a 100-mm Visual Analog Scale (VAS), including Hunger, Desire to Eat, Fullness, and Prospective Food Consumption. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores on Hunger, Desire to Eat, and Prospective Food Consumption indicate greater appetite drive and poorer satiety; higher scores on Fullness indicate greater satiety (better outcome).
Composite Appetite Score Positive Maximum Response | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Maximum positive change from fasting baseline in the Composite Appetite Score, calculated as the average of standardized 100-mm Visual Analog Scale (VAS) ratings for Hunger, Desire to Eat, Fullness, and Prospective Food Consumption. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher values for Hunger, Desire to Eat, and Prospective Food Consumption reflect increased appetite, while higher values for Fullness reflect enhanced satiety; the composite score is interpreted based on the net direction of these opposing components (better outcome).
Individual Appetite Visual Analog Scale (VAS) Ratings Positive Maximum Response | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Maximum positive deviation from fasting baseline in individual appetite-related sensations measured using a 100-mm Visual Analog Scale (VAS) for Hunger, Desire to Eat, Fullness, and Prospective Food Consumption. The scale ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores on Hunger, Desire to Eat, and Prospective Food Consumption represent greater appetite and poorer satiety; higher scores on Fullness represent stronger satiety (better outcome) .
Energy Composite Score Net Incremental Area Under the Curve (niAUC) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Net incremental area under the curve (niAUC) from 0 to 120 minutes for the Energy Composite Score, derived as the mean of three 100-mm Visual Analog Scale (VAS) items: Energy, Vigor, and Pep. Each VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores indicate greater perceived energy levels and are interpreted as a better outcome.
Energy Composite Score Positive Maximum Response | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Maximum positive change from fasting baseline in the Energy Composite Score, calculated as the average of three 100-mm Visual Analog Scale (VAS) ratings: Energy, Vigor, and Pep. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores reflect greater increases in subjective energy and are considered a better outcome.
Fatigue Composite Score Net Incremental Area Under the Curve (niAUC) | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Net incremental area under the curve (niAUC) from 0 to 120 minutes for the Fatigue Composite Score, calculated as the mean of three 100-mm Visual Analog Scale (VAS) items: Fatigue, Exhaustion, and Worn-out. Each VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores indicate greater perceived fatigue and are interpreted as a worse outcome.
Fatigue Composite Score Positive Maximum Response | Baseline (Visit 2, Day 1): t=0 to t=120 minutes
  Maximum positive change from fasting baseline in the Fatigue Composite Score, derived from the average of three 100-mm Visual Analog Scale (VAS) ratings: Fatigue, Exhaustion, and Worn-out. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores reflect greater increases in perceived fatigue and are considered a worse outcome.
Waist Circumference (WC) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in in-clinic measured Waist Circumference from Baseline to the End of the Study.
Hip Circumference (HC) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in in-clinic measured Hip Circumference from Baseline to the End of the Study.
Waist-to-Hip Ratio (WHR) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in calculated Waist-to-Hip Ratio (WC/HC) from Baseline to the End of the Study.
Lean Mass | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in total and regional (arms, legs, trunk) lean mass, measured via Dual-energy X-ray Absorptiometry (DXA), from Baseline to the End of the Study.
Fat Mass | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in total and regional (arms, legs, trunk) fat mass, measured via DXA, from Baseline to the End of the Study.
Fat-Free Mass | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in total fat-free mass, measured via DXA, from Baseline to the End of the Study.
Visceral Adipose Tissue (VAT) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in abdominal visceral fat mass and volume, measured via DXA, from Baseline to the End of the Study.
Fasting Plasma Glucose | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in fasting plasma glucose levels from Baseline to the End of the Study.
Fasting Plasma Insulin | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in fasting plasma insulin levels from Baseline to the End of the Study.
Glycated Hemoglobin (HbA1c) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in Glycated Hemoglobin (HbA1c) levels from Baseline to the End of the Study.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in HOMA-IR calculated from fasting glucose and insulin levels from Baseline to the End of the Study.
Fasting Plasma Leptin | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in fasting plasma leptin levels from Baseline to the End of the Study.
Postprandial Glucose niAUC (0-120 min) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in postprandial glucose niAUC (0-120 min) response to an MTT from Baseline to the End of the Study.
Postprandial Glucose Cmax | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in postprandial glucose Cmax response to an MTT from Baseline to the End of the Study.
Postprandial Glucose Tmax | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in postprandial glucose Tmax response to an MTT from Baseline to the End of the Study.
Postprandial Appetite Visual Analog Scale (VAS) Net Incremental Area Under the Curve (niAUC; 0-120 minutes) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change from baseline to end of study in the net incremental area under the curve (niAUC) over 0 to 120 minutes for postprandial appetite ratings measured using a 100-mm Visual Analog Scale (VAS), including Hunger, Desire to Eat, Fullness, and Prospective Food Consumption. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores on Hunger, Desire to Eat, and Prospective Food Consumption indicate greater appetite drive and poorer satiety ; higher scores on Fullness indicate greater satiety (better outcome).
Postprandial Appetite Visual Analog Scale (VAS) Positive Maximum Response | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change from baseline to end of study in the positive maximum response (maximum increase from fasting value) of postprandial appetite ratings measured using a 100-mm Visual Analog Scale (VAS), including Hunger, Desire to Eat, Fullness, and Prospective Food Consumption. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores on Hunger, Desire to Eat, and Prospective Food Consumption indicate greater appetite drive and poorer satiety; higher scores on Fullness indicate greater satiety (better outcome).
Postprandial Energy Visual Analog Scale (VAS) Net Incremental Area Under the Curve (niAUC; 0-120 min) | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change from baseline to end of study in the net incremental area under the curve (niAUC) over 0-120 minutes for postprandial energy-related ratings measured using a 100-mm Visual Analog Scale (VAS), including Energy, Vigor, and Pep. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher niAUC values indicate greater postprandial energy enhancement and are interpreted as a better outcome.
Postprandial Energy Visual Analog Scale (VAS) Positive Maximum Response | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change from baseline (Week 0) to end of study (Week 12) in the incremental peak response (defined as the maximum increase from the pre-meal fasting value) for postprandial energy-related ratings. Ratings are assessed using a 100-mm Visual Analog Scale (VAS) for three items: Energy, Vigor, and Pep. The VAS ranges from 0 mm ("not at all") to 100 mm ("extremely"). Higher scores represent a greater maximal increase in perceived energy levels, indicating a better outcome.
Profile of Mood States -2 (POMS-2) Total and Component Scores | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change from baseline to end of study in the POMS-2 Total Mood Disturbance (TMD) score and six component subscale scores: Anger-Hostility, Confusion-Bewilderment, Depression-Dejection, Fatigue-Inertia, Tension-Anxiety, and Vigor-Activity. The POMS-2 is a validated 65-item self-report questionnaire rated on a 5-point Likert scale (0 = "Not at all" to 4 = "Extremely"). The TMD score is calculated by summing the scores of the five negative mood subscales and subtracting the Vigor-Activity score. Higher TMD and negative subscale scores reflect greater emotional distress (worse outcome), while higher Vigor-Activity scores reflect increased energy and well-being (better outcome).

OTHER OUTCOMES:
Number of participants with abnormal Clinical Chemistry Panel (CMP) tests result | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Number of participants with CMP analyte values (including albumin, alkaline phosphatase, total bilirubin, direct bilirubin, calcium, chloride, creatinine, BUN, potassium, AST, ALT, sodium, total protein, CO2, and osmolality) that are outside the reference range and considered clinically significant by the investigator.
Number of participants with abnormal Complete Blood Count (CBC) tests result | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Number of participants with CBC analyte values (including WBC, RBC, hemoglobin concentration, hematocrit, MCV, MCH, MCHC, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelet count) that are outside the reference range and considered clinically significant by the investigator.
Blood Pressure | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in resting systolic blood pressure and diastolic blood pressure from Baseline to the End of the Study.
Heart Rate | Baseline (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Change in resting heart rate from Baseline to the End of the Study.
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Start of study product consumption (Visit 2, Week 0, Day 1) to End of the Study (Visit 3, Week 12, Day 84)
  Incidence, type, severity, and relationship to the study product of AEs and SAEs occurring during the chronic phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Merieux NutriSciences, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderssen S, Holme I, Urdal P, Hjermann I. Diet and exercise intervention have favourable effects on blood pressure in mild hypertensives: the Oslo Diet and Exercise Study (ODES). Blood Press. 1995 Nov;4(6):343-9. doi: 10.3109/08037059509077619. PMID 8746601
- [Background] Herrera-Acosta J, Reyes PA, Lopez Manay G, Padilla L, Cerdas Calderon M, Ruiz A, Perez Grovas H. [Inhibition of prostaglandin synthesis suppresses the renal functional reserve in patients with lupus nephropathy]. Rev Invest Clin. 1987 Apr-Jun;39(2):107-14. No abstract available. Spanish. PMID 3310165
- [Background] Zhang H, Wei J, Xue R, Wu JD, Zhao W, Wang ZZ, Wang SK, Zhou ZX, Song DQ, Wang YM, Pan HN, Kong WJ, Jiang JD. Berberine lowers blood glucose in type 2 diabetes mellitus patients through increasing insulin receptor expression. Metabolism. 2010 Feb;59(2):285-92. doi: 10.1016/j.metabol.2009.07.029. Epub 2009 Oct 1. PMID 19800084
- [Background] Chan M, Qin Z, Man SC, Lam M, Lai WH, Ng RMK, Lee CK, Wong TL, Lee EHM, Wong HK, Feng Y, Liu L, Han F, Chen EYH, Zhang ZJ. Adjunctive berberine reduces antipsychotic-associated weight gain and metabolic syndrome in patients with schizophrenia: a randomized controlled trial. Psychiatry Clin Neurosci. 2022 Mar;76(3):77-85. doi: 10.1111/pcn.13323. Epub 2022 Jan 18. PMID 34931749